CLINICAL TRIAL: NCT04380467
Title: Impact of Vitamin D Supplementation on Vascular Function, Vascular Structure and Immune Regulation in Patients With Chronic Kidney Disease and Low Vitamin D Levels - A Pilot Randomised Trial
Brief Title: Vitamin D Supplementation in CKD - Vascular Function, Structure and Immune Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15.0236
Record Dates: First submitted 2016-07-19; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Atherosclerosis; Chronic Kidney Disease
Keywords: Vitamin D; Cholecalciferol; Chronic Kidney Disease; Cardiovascular Disease; Atherosclerosis; Flow Mediated Dilatation; Carotid Intima Media Thickness; CD4+CD28null T lymphocyte; Regulatory T lymphocyte
MeSH Terms: conditions — Atherosclerosis; Renal Insufficiency, Chronic; Cardiovascular Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D Group (Experimental): Six doses of cholecalciferol 100,000units (5x aviticol 20,000units capsules) administered monthly over 20 weeks.
  Interventions: Dietary Supplement: Vitamin D (cholecalciferol)
- Control (No Intervention): No vitamin D given

INTERVENTIONS:
Dietary Supplement: Vitamin D (cholecalciferol) — (aviticol) 5x 20,000unit capsules administered monthly over 20 weeks
  Arms: Vitamin D Group

SUMMARY:
A pilot study to assess feasibility of methods of an observer-blinded randomised controlled trial of the effect of vitamin D supplementation in Chronic Kidney Disease and low vitamin D levels on markers of vascular function (Flow Mediated Dilatation of Brachial Artery), vascular structure (Carotid Intima Media Thickness) and Immune Regulation (frequencies of CD4+CD28null T lymphocytes ad Regulatory T lymphocytes).

DETAILED DESCRIPTION:
The study is a single (observer) blinded feasibility pilot randomised study. Study subjects will be recruited from clinics run by St George's Hospital Renal Department and randomised to treatment arm or no treatment arm.

In treatment arm, six doses of vitamin D tablets (cholecalciferol 100,000 IU, five capsules total) will be administered on weeks 0, 4, 8, 12, 16 and 20. In the no-treatment arm the participants receive no cholecalciferol. Participants will have serum calcium levels measured at week 12.

All participants will undergo estimation of endothelial function, carotid intima-media thickness, CD4+CD28null and regulatory T cell frequency in week 0 and week 26. The observer will be blinded to whether the patient is in the treatment or no-treatment arm whilst the following tests are performed:

1. Measurement of Brachial Artery Flow Mediated Dilatation
2. Measurement of Carotid Intima Media Thickness
3. Quantification of CD4+CD28null and regulatory T cell frequency

The pilot study will assess feasibility of the study methods.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. Calcium < 2.58mmol/l
3. On an ACE inhibitor/ARB
4. Vitamin D <75nmol/l
5. eGFR 15- 60ml/min/1.73m2 and stable
6. Informed consent to participate

Exclusion Criteria:

1. Patients already on Vitamin D or calcium supplementation
2. Patients with known malignancies
3. Patients with autoimmune conditions
4. Patients with heart failure (ejection fraction <40%, Plasma NT pro-BNP>500pg/ml)
5. Patients with active infection
6. Rapidly deteriorating renal function
7. Recent Acute coronary syndrome or cerebro-vascular event (within the last 6 months)
8. Uncontrolled hypertension (BP>160 systolic)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 3 months
  Percentage of patients recruited from those eligible for the study.
Retention rate | 6 months
  Percentage of patients recruited who completed the follow up investigations
Acceptability to patients of randomisation procedures | 6 months
  Acceptability as assessed by quantitative and qualitative analysis of Participant Experience Survey
Randomisation procedure | 6 months
  Comparison of baseline indices of two patient groups
Maintenance of single (observer) blinding | 6 months
  Incidences of unblinding of study investigator
Adherence to vitamin D supplementation | 6 months
  Subjective adherence as assessed by Participant Experience Survey and biochemical correlation by comparison of follow up vitamin D levels

SECONDARY OUTCOMES:
Witnessed change in FMD between treated and untreated subjects | 6 months
  Flow Mediated Dilatation
Witnessed change in CIMT between treated and untreated subjects | 6 months
  Carotid Intima Media Thickness
Witnessed change in T lymphocyte subset frequency between treated and untreated subjects | 6 months
  CD4+CD28null T lymphocytes and Regulatory T cells as determined by flow cytometry of whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Debasish Banarjee, Principal Investigator — St Georges University NHS Foundation Trust
Locations (1):
- Debasish Banerjee, London, Tooting, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided